CLINICAL TRIAL: NCT07082868
Title: A Phase Ib Trial With Dose Expansion of Epcoritamab in Combination With Ibrutinib in Refractory/Recurrent CNS Lymphoma (EIFEL-Trial)
Brief Title: A Study of Epcoritamab and Ibrutinib in People With Central Nervous System Lymphoma (CNSL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-032
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL); Primary Central Nervous System Lymphoma; Relapsed Primary Central Nervous System Lymphoma; Refractory Primary Central Nervous System Lymphoma; Central Nervous System Lymphoma; Secondary Central Nervous System Lymphoma; Secondary Central Nervous System Lymphoma (SCNSL)
Keywords: Primary Central Nervous System Lymphoma; PCNSL; Relapsed Primary Central Nervous Lymphoma; Refractory Primary Central Nervous Lymphoma; Central Nervous System Lymphoma; Secondary Central Nervous System Lymphoma; SCNSL; epcoritamab; ibrutinib; 25-032; Memorial Sloan Kettering Cancer Center
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Relapsed or refractory PCNSL (n=6)
  Interventions: Drug: ibrutinib; Drug: Epcoritamab
- Cohort B1 (Experimental): Relapsed or refractory PCNSL (n=10)
  Interventions: Drug: ibrutinib; Drug: Epcoritamab
- Cohort B2 (Experimental): Relapsed or refractory PCNSL (n=10)
  Interventions: Drug: ibrutinib; Drug: Epcoritamab

INTERVENTIONS:
Drug: ibrutinib — Ibrutinib should be self-administered daily by the participant and should be taken at approximately the same time each day
Drug: Epcoritamab — Epcoritamab will be administered at the study site clinic, as a SC injection

SUMMARY:
The purpose of this study is to find out whether the combination of epcoritamab and ibrutinib is a safe treatment approach that causes few or mild side effects in people with relapsed/refractory primary central nervous system lymphoma (PCNSL) or secondary central nervous system lymphoma (SCNSL).

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years of age on the day of consenting to the study.
* Histologically documented DLBCL at enrolling institution (biopsy or CSF samples in PCNSL; biopsy of CNS or non-CNS sample in SCNSL)
* Participants must have an ECOG performance status of 0, 1, or 2.
* Participants must have adequate bone marrow and organ function shown by:

  * Absolute neutrophil count (ANC) ≥ 1 x 109/L
  * Platelets ≥ 75 x 109/L and no platelet transfusion within the past 21 days prior to study consent
  * Hemoglobin (Hgb) ≥ 8 g/dL and no red blood cell (RBC) transfusion within the past 21 days prior to study consent
  * International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal (unless receiving anticoagulation)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal
  * Serum bilirubin ≤ 1.5 times the upper limit of normal; or total bilirubin ≤ 3 times the upper limit of normal with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome.
  * Creatinine clearance (CLCr) ≥ 30 ml/min (based on the following formular Creatinine clearance= ((140-age)*wt)/(creatinine*72); multiply by 0.85 for women)
* Women of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 30 days after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 3 months after the last dose
* Female subjects of childbearing potential must have a negative serum pregnancy test upon study entry. See section on Pregnancy and Reproduction.

  * Patients must be able to tolerate MRI/CT scans.
  * Due to the nature of this disease, we will allow patients with impaired decision-making ability to enroll into all cohorts.

Exclusion Criteria:

* Newly diagnosed PCNSLs or SCNSLs and patients with non-CNS disease are excluded.
* Patients with existing chronic moderate and severe hepatic impairment (Child-Pugh class B or C) are excluded
* Patient is concurrently using other approved or investigational antineoplastic agents.
* Patient has an active concurrent malignancy requiring active therapy
* Patient has received chemotherapy, monoclonal antibodies or targeted anticancer therapy ≤ 4 weeks or 5 half-lives, whichever is shorter, or 6 weeks for nitrosourea or mitomycin-C prior to starting the study drug, or the patient has not recovered from the side effects of such therapy.
* Patient has received external beam radiation therapy to the CNS within 21 days of the first dose of the study drug.
* Patient requires more than 8 mg of dexamethasone daily or the equivalent
* Patient is using warfarin or any other warfarin-derivative anticoagulant or vitamin K antagonists. Patients must be off warfarin-derivative anticoagulants for at least seven days prior to starting the study drug. Low molecular weight heparin is allowed. Patients with congenital bleeding diathesis are excluded.
* Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or starfruit for at least 3 days prior to Cycle 1 Day 1
* Patient is taking a drug known to be a moderate or strong inhibitor or inducers of the P450 isoenzyme CYP3A. Participants must be off P450/CYP3A inhibitors and inducers for at least 5 half-lives or at least two weeks, whichever is shorter, prior to starting the study drug.
* Patient is using systemic immunosuppressant therapy, including cyclosporine A, tacrolimus, sirolimus, and other such medications, or chronic administration of > 5 mg/day of prednisone or the equivalent (for more than 12 months). Participants must be off of immunosuppressant therapy for at least 28 days prior to the first dose of the study drug.
* Patient has significant abnormalities on screening electrocardiogram (EKG) and active and significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, hypertension, valvular disease, pericarditis, or myocardial infarction within 6 months of screening
* Patient has an ejection fraction of <50%
* Patient has a known bleeding diathesis (e.g. von Willebrand's disease) or hemophilia.
* Patient is documented to have human immunodeficiency virus (HIV) infection.
* Patient is documented to have a history of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests.
* Patient is known to have an uncontrolled active systemic infection.
* Patient is unable to swallow capsules or has a disease or condition significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, or complete bowel obstruction.
* Patient has a life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject's safety or put the study outcomes at undue risk.
* Patient has not received vaccination with live vaccines within 28 days prior to first dose of study drug or is expected to need any live vaccination during study participation including at least 3 months following the last dose of study treatment. Note: COVID-19 non-replicating adenoviral vaccines are permitted with a minimum period of 3 days between the vaccine and a dose of study drug. It is highly recommended that every patient enrolled onto this trial has updated vaccination status (e.g. flu, hepatitis, polio, pertussis, tetanus; when is doubt please contact the PI or side-PI).
* Women who are pregnant or nursing (lactating), where pregnancy is defined as a state of a female after conception until the termination of gestation, confirmed by a positive serum hCG laboratory test of > 5 mIU/mL

Pregnancy and Reproduction

Women:

* Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy with or without hysterectomy at least six weeks prior to enrollment in the study. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up of hormone level assessment is she considered not of childbearing potential.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during study treatment and for 4 months after study discontinuation. Highly effective contraception is defined as either

  * True abstinence: When this is the line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Sterilization: Surgical bilateral oophorectomy, with or without hysterectomy, or tubal ligation at least six weeks prior to study enrollment.
  * Male partner sterilization (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female patients participating in the study, the vasectomized male partner should be the sole partner for that patient.
  * Use of a combination of any two of the following:
* Placement of an intrauterine device (IUD) or intrauterine system (IUS)
* Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical vault caps) with spermicidal form/gel/film/cream/vaginal suppository
* Women of child-bearing potential must have one negative serum pregnancy tests at screening
* In addition to having a negative pregnancy test confirmed at screening, all female participants of child bearing potential must have a negative pregnancy test confirmed within 48 hours prior to dosing with the study drug.

Men:

* Fertile males, defined as all male subjects physiologically capable of conceiving offspring, must use a condom during study treatment and for 4 months after study discontinuation and should not father a child in this period.
* Female partner of a male study subject should use a highly effective method of contraception while the male partner is receiving the study agent and for 4 months after the final dose of the study therapy.

Inclusion of women, minorities or other underrepresented populations

* Ibrutinib and epcoritamab are not known to differentially affect subpopulations, including women, minorities, or other underrepresented groups. The eligibility and exclusion criteria are not expected to differentially impact recruitment or retention of these subpopulations.

Covid-19 eligibility criteria

Subject has no known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. If a subject has signs/symptoms suggestive of SARS-CoV-2 infection or have had recent known exposure to someone with SARS-CoV-2 infection, the subject must have a negative molecular (e.g., PCR) test, or 2 negative antigen test results at least 24 hours apart, to rule out SARS-CoV-2 infection.

Subjects who do not meet SARS-CoV-2 infection eligibility criteria must be screen failed and may only rescreen after they meet the following SARS-CoV-2 infection viral clearance criteria:

* No signs/symptoms suggestive of active SARS-CoV-2 infection
* Negative molecular (e.g., PCR) result or 2 negative antigen test results at least 24 hours apart

Given the ongoing COVID-19 pandemic, selected non-live vaccines (e.g. mRNA, non-replicating viral vector, protein subunit, etc.) to prevent SARS-CoV-2 infections may be administered during screening or the treatment period, as long as components of the vaccine are not contraindicated. COVID-19 vaccines are permitted and strongly recommended.

The decision to receive a locally available vaccine should be based on local guidance and an individual discussion between the treating physician and the subject.

The potential impact of epcoritamab on SARS-CoV-2 vaccination is unknown. Therefore, study drug should be administered as follows:

* The first dose of study drug, when possible, is preferred to be given at least 14 days from SARS-CoV-2 vaccine administration.
* A minimum period of 3 days must occur between the administration of an appropriate COVID-19 vaccine and the administration od epcoritamab (to avoid overlapping AEs).

Note: The above guidance applies to all SARS-CoV-2 vaccine doses given as part of the complete vaccination course.

These recommendations may be subject to change based on the evolving knowledge around the use of SARS-Cov-2 vaccines in subjects with recurrent/refractory DLBCL or cFL and as more data are collected in real-world scenarios and clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Number of dose limiting toxicities/DLTs | 8 weeks
  Cohort A - To determine the safety and tolerability of epcoritamab in combination with ibrutinib in CNS lymphoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grommes, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org